CLINICAL TRIAL: NCT03295994
Title: Operative Versus Non-Operative Treatment for Atraumatic Rotator Cuff Tears: A Multicenter Randomized Controlled Pragmatic Trial
Brief Title: Operative Versus Non-Operative Treatment for Atraumatic Rotator Cuff Tears
Acronym: ARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Nitin Jain, Professor of Physical Medicine & Rehabilitation, and Orthopaedics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 171863; 1605-35413 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Tear
Keywords: arthroscopy; physical therapy; rehabilitation; surgery; rotator cuff tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Operative (Active Comparator): surgery + post-operative physical therapy
  Interventions: Procedure: Operative
- Non-Operative (Active Comparator): non-operative physical therapy
  Interventions: Procedure: Non-Operative

INTERVENTIONS:
Procedure: Operative — Arthroscopic rotator cuff surgery followed by physical therapy.
  Arms: Operative
Procedure: Non-Operative — Physical therapy (without surgery).
  Arms: Non-Operative

SUMMARY:
Rotator cuff tears are one of the most common reasons to seek musculoskeletal care in the United States and one of the fastest growing ambulatory surgery procedures. However, data on comparison of operative versus non-operative treatment is lacking and urgently needed.

DETAILED DESCRIPTION:
This is non-blinded, randomized controlled trial. Patients will be randomly assigned to either an operative or non-operative course of treatment and will be followed for 12 months from baseline.

Aim 1: To compare pain and function in patients undergoing operative versus non-operative treatment of atraumatic rotator cuff tears at 12 months of follow-up

Aim 2: To assess effects of rotator cuff tear size and age on comparative outcomes of operative versus non-operative treatments for atraumatic rotator cuff tears

5U34AR069201-02 NIH grant funded the preparatory work for the trial but not the trial itself.

ELIGIBILITY:
Inclusion Criteria:

* Aged =>40 years to <85 years
* Shoulder pain and/or loss of range of active motion, strength or function
* MRI-confirmed partial- or full-thickness supraspinatus and/or infraspinatus tear of 4cm or less in longitudinal dimension
* Medically fit for surgery, defined as Category I-III per American Society of Anesthesiologists (ASA) Physical Status Classification
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Primary diagnosis is something other than a rotator cuff tear
* History (in last 2 years) of shoulder fracture involving the humeral head on affected side
* Previous rotator cuff surgery on affected side
* Isolated subscapularis &/or teres minor tear on affected side
* Acute rotator cuff tear caused by a severe trauma
* Shoulder used as a weight-bearing joint
* Contraindication to MRI (claustrophobia, pacemaker, pregnancy, shoulder implant, etc.)
* Glenohumeral osteoarthritis on xrays/MRI, as determined by recruiting MD
* Grade 4 fatty infiltration of rotator cuff (any tendons)
* Candidate for shoulder arthroplasty at baseline
* Non-English speaking

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain & Disability Index (SPADI) | Study participants will be followed for 12 months
  SPADI is a composite pain and function measure. The scale range is from 0 to 100, with 0 being best, and 100 being worst.

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) | Study participants will be followed for 12 months
  ASES is a pain and activity of daily living questionnaire. The range is from 0 to 100, with 0 being worst, and 100 being best.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Jain, MD,MSPH, Principal Investigator — University of Michigan
Locations (19):
- United States (19):
  - University of California - San Francisco (UCSF), San Francisco, California
  - Western Orthopaedics, Denver, Colorado
  - University of Colorado - Denver, Denver, Colorado
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Orthopedic Institute, Sioux Falls, South Dakota
  - Ortho Tennessee - Knoxville Orthopedic Clinic, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Ortho Virginia, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jain NB, Ayers GD, Koudelkova H, Archer KR, Dickinson R, Richardson B, Derryberry M, Kuhn JE; ARC Trial Group. Operative vs Nonoperative Treatment for Atraumatic Rotator Cuff Tears: A Trial Protocol for the Arthroscopic Rotator Cuff Pragmatic Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e199050. doi: 10.1001/jamanetworkopen.2019.9050. PMID 31397866
- See also: ARC Trial website — https://shoulderstudy.org/studies/arc-trial/